CLINICAL TRIAL: NCT06274580
Title: Endovascular vs Conservative Treatment in Patients With Chronic Subdural Hematomas and Mild Symptoms: a Multicentre Randomized Trial
Brief Title: Endovascular vs Conservative Treatment in Patients With Chronic Subdural Hematomas and Mild Symptoms
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ospedale Policlinico San Martino (Other)
Responsible Party: Principal Investigator, Castellan, MD, Ospedale Policlinico San Martino
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5916
Record Dates: First submitted 2024-02-06; First posted 2024-02-23 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Subdural Hematoma, Chronic
Keywords: subdural hematoma; chronic; embolization; middle meningeal artery
MeSH Terms: conditions — Hematoma, Subdural, Chronic; Hematoma, Subdural; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Embolization of the middle meningeal artery (Experimental): Endovascular treatment of chronic subdural hematoma
  Interventions: Device: embolization of the middle meningeal artery
- standard of care (No Intervention): control group will managed according to the current standard of care with "wait and see" approach and best medical treatment

INTERVENTIONS:
Device: embolization of the middle meningeal artery — Embolization of the MMA is occluded with PVA particles or liquid embolizing materials
  Arms: Embolization of the middle meningeal artery

SUMMARY:
Embotrial-1 is an Italian multicenter prospective randomized clinical trial with open-label treatment and blinded outcome assessment (PROBE) to assess the superiority of MMA embolization compared to conservative treatment. The intervention group is MMA embolization and comparator control group is the conservative management with best medical treatment. Patients are randomized 1:1.

DETAILED DESCRIPTION:
Patients randomized to the experimental arm will submit to cerebral angiography and bilateral MMA embolization of the cSHD, even if it is located to only one side. The ipsilateral MMA embolization of the cSDH is allowed when the endovascular procedure cannot be performed on both sides. Patients are preferably under monitored local anesthesia or alternatively under conscious sedation or general anesthesia. Briefly, through femoral or radial artery access a standard 5 French diagnostic catheter is placed in the proximal external carotid artery and a digital subtraction angiography (DSA) is performed. Then, a microcatheter is advanced selectively under roadmap guidance into the main trunk of MMA, and superselective angiography is performed to evaluate for potentially dangerous anastomoses between MMA and ophthalmic or petrous branches prior to embolization. After collateral vessels are excluded, the MMA is occluded with PVA particles or liquid embolizing materials . The successful embolization is defined as that both frontal and parietal branch of MMA are selectively occluded and for this purpose, the microcatheter should be placed as distally as possible. It is recommended to ensure embolic materials penetrating into the capillary network of the dura to be permanently blocked. Patients randomized to the conservative arm will be clinmically monitored and eventually receive a best supportive care according to the local practice.

The trial is powered to assess superiority. When assuming the event rate of 1% in intervention group and 10% event rate in the control group, with a power of 85% and two-sided alpha of 0.05, allowing for 10% drop-outs, the estimated sample size is 300 patients in total.

The safety and efficacy interim analysis will be planned when half of the target sample (150 patients) completed 6 months follow-up. The enrollment will be stopped if the futility assessment based on estimated conditional power will be <70%.

All patient data is registered in the electronic data capture software REDCap. This worldwide online system allows built-in logical checks and validations to promote data quality. All clinical data are entered via an encrypted connection, are anonymized, and fulfill the demands for data protection. All data entries and changes are logged in REDCap and meet the Good Clinical Practice (GCP) requirements for the use of the electronic case report form (eCRF) in medical trials. Trial coordinators, data managers and the investigators will be introduced to the platform and trained in data entry during the initial kick-of meeting prior to recruitment of the first patient. Trial staff will be provided with a personal ID.

Currently, 6 centers in Italy have been identified for the study. All the clinical investigators are board-certified and have renowned expertise in neurosurgery, neuroradiology and endovascular interventions.

ELIGIBILITY:
Inclusion Criteria:

* No neurological deficits (Markwalder score ≤1);
* Unilateral or bilateral cSDH;
* Subdural Hematoma width ≤ 20 mm; midline shift ≤ 7mm;
* Independent functional status with mRS score ≤ 2 prior to symptom onset;
* Likely compliance of the participant in attending follow-up examination.

Exclusion Criteria:

* Radiological evidence of an acute or subacute subdural hematoma, subarachnoid hemorrhage, intracerebral hematoma or epidural hematoma;
* Contraindications to angiography (end stage chronic renal disease, any sign of anatomical variations that could make MMA embolization unsafe, pregnancy);
* Life expectancy < 1 year;
* Patients with any kind of ventricular derivation catheter.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Rate of incomplete hematoma resolution or surgical rescue | 6 months
  Incomplete hematoma resolution is defined as a reduction of the cSDH thickness ≤50% at follow-up compared to the hematoma thickness measured at the time of randomization. Surgical rescue is intended as hematoma removal for relief of symptoms (mRS≥3 and Markwalder scale≥2) that develope with progressive growth of the cSDH

SECONDARY OUTCOMES:
treatment complication | 30 days
  Procedure related complication during or 30 days after MMA embolization
treatment successful | periprocedural
  Successful embolization rate of the target vessels based on angiographic findings

CONTACTS AND LOCATIONS:
Overall Officials: Lucio Castellan, MD, Principal Investigator — Ospedale Policlinico San Martino

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Santarius T, Kirkpatrick PJ, Ganesan D, Chia HL, Jalloh I, Smielewski P, Richards HK, Marcus H, Parker RA, Price SJ, Kirollos RW, Pickard JD, Hutchinson PJ. Use of drains versus no drains after burr-hole evacuation of chronic subdural haematoma: a randomised controlled trial. Lancet. 2009 Sep 26;374(9695):1067-73. doi: 10.1016/S0140-6736(09)61115-6. PMID 19782872
- [Result] Kim HC, Ko JH, Yoo DS, Lee SK. Spontaneous Resolution of Chronic Subdural Hematoma : Close Observation as a Treatment Strategy. J Korean Neurosurg Soc. 2016 Nov;59(6):628-636. doi: 10.3340/jkns.2016.59.6.628. Epub 2016 Oct 24. PMID 27847578
- [Result] Rojas-Villabona A, Mohamed S, Kennion O, Padmanabhan R, Siddiqui A, Prasad M, Mukerji N. A systematic review of middle meningeal artery embolization for minimally symptomatic chronic subdural haematomas that do not require immediate evacuation. Brain Spine. 2023 Sep 6;3:102672. doi: 10.1016/j.bas.2023.102672. eCollection 2023. PMID 38021007
- [Result] Akamatsu Y, Kashimura H, Kojima D, Yoshida J, Chika K, Komoribayashi N, Fujiwara S, Ogasawara K. Correlation Between Low-Density Hematoma at 1-Week Post-Middle Meningeal Artery Embolization and Rapid Resolution of Chronic Subdural Hematoma. World Neurosurg. 2024 Jan;181:e1088-e1092. doi: 10.1016/j.wneu.2023.11.045. Epub 2023 Nov 17. PMID 37979682
- [Result] Omura Y, Ishiguro T. Middle meningeal artery embolization for chronic subdural hematoma: a systematic review. Front Neurol. 2023 Oct 10;14:1259647. doi: 10.3389/fneur.2023.1259647. eCollection 2023. PMID 37881312
- [Derived] Salsano G, Fiaschi P, Laura G, Sonia M, Fontana V, Boni L, Zona G, Castellan L. Endovascular vs conservative treatment in patients with chronic subdural hematomas and mild symptoms: a study protocol for a multicenter randomized controlled trial (EMBOTRIAL-1). Trials. 2025 Nov 18;26(1):517. doi: 10.1186/s13063-025-09131-y. PMID 41254694